CLINICAL TRIAL: NCT07231744
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of STLX-2012 in Healthy Volunteers
Brief Title: Study of STLX-2012 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stelexis BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STLX-2012-001
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STLX-2012 (Experimental): Single ascending doses of STLX-2012
  Interventions: Drug: STLX-2012
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: STLX-2012 — STLX-2012 IV
  Arms: STLX-2012
Other: Placebo — Placebo arm
  Arms: Placebo

SUMMARY:
The purpose of this research is to establish the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of a single IV dose of STLX-2012.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18-55 years old, inclusive, at Screening.
* Body mass index of 18-32 kg/m^2, inclusive
* Healthy as determined by the investigator
* Adequate hepatic and renal function
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Male participants and females of childbearing potential must agree to use an effective method of contraception for 30 days after the last dose of STLX-2012

Exclusion Criteria:

* Pregnant or lactating female.
* Positive urine drug screen or alcohol breath test
* Neutropenia, defined as neutrophil count <2.0 x 10^9/L
* History of allergic reaction requiring treatment or anaphylactic reactions to any therapeutic drug.
* Previous treatment with an IL-1RAP monoclonal antibody
* History of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, inflammatory, or allergic disease (excluding mild seasonal allergies)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs, graded according to the NCI CTCAE Version 6.0 | 56 days

SECONDARY OUTCOMES:
Pharmacokinetics of STLX-2012: area under the plasma concentration-time curve (AUC) | Day 1 - 29
Pharmacokinetics of STLX-2012: maximum observed serum concentration (Cmax) | Day 1 - 29
Pharmacokinetics of STLX-2012: time corresponding to the occurrence of Cmax (Tmax) | Day 1 - 29
Pharmacokinetics of STLX-2012: apparent terminal elimination half-life (t½) | Day 1 - 29
Pharmacokinetics of STLX-2012: Clearance (CL) | Day 1 - 29
Pharmacokinetics of STLX-2012: Volume of distribution (Vd) | Day 1 - 29

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Brisbane, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No plans or process in place for sharing IPD